CLINICAL TRIAL: NCT00875589
Title: Eye-movement Recordings in the Diagnosis of Traumatic Brain Injury
Brief Title: Eye Movement Recordings in the Diagnosis of Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: B6403-R
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Eye movement recording
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Control subjects with no Mild Traumatic Brain Injury (MTBI) and no Post-Traumatic Stress Disorder (PTSD)
- MTBI: Subject with a diagnosis for Mild Traumatic Brain Injury (MTBI)

SUMMARY:
The study investigates whether the use of eye movement recordings can provide a reliable diagnostic of previously undiagnosed mild traumatic brain injury (blast and impact) in Operations Enduring Freedom or Iraqi Freedom (OIF/OEF) veterans.

DETAILED DESCRIPTION:
Eye movements are recorded for Operations Enduring Freedom or Iraqi Freedom (OIF/OEF) veterans with mild traumatic brain injury (mTBI) and compared to the eye movements of those without mTBI. By analyzing and characterizing the differences between the two groups, a diagnostic measure of mTBI through the use of eye movements can be developed.

ELIGIBILITY:
Inclusion Criteria:

* OIF/OEF Veteran;
* Neuropsych diagnosis of MTBI

Exclusion Criteria:

* chronically abusing alcohol or illicit drugs.
* uncorrected vision prevents subject from effectively viewing the stimuli, unless they can wear contact lenses during the recording session.
* inability to make normal eye movements (i.e.: saccades, smooth pursuit) required by study paradigms. Note: Deficit can be caused by taking medications that can potentially affect eye movements or any neurological condition that can interfere with making normal eye movement.
* psychological or psychiatric conditions that preclude sustained concentration or ability to perform the tasks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult betwenn 18 and 55 years old with and without a diagnosis of MTBI
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Jacobs, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Controls: Control Group - subjects with no Mild Traumatic Brain Injury (MTBI)
- MTBI: MTBI Group - subjects with diagnosed Mild Traumatic Brain Injury (MTBI)
Period: Overall Study
Arm/Group | Controls | MTBI
Started | 15 | 11
Completed | 15 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Controls | MTBI | Total
Number analyzed (Participants) | 15 | 11 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 11 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Stability of Fixation
Description: The ability to keep eye position fixed on a visual target, measured by the distance between the target and eye fixation point averaged over 20 sec.
Time Frame: During eye movement recording session (20 sec).
Population: Although there were 15 participants in the Control arm, data were only analyzed for a cohort of 11 that were age-matched to the MTBI arm participants.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Controls | MTBI
Number analyzed (Participants) | 11 | 11
degrees | 0.8 (0.01) | 1.1 (0.1)

ADVERSE EVENTS:
Arm/Group | Controls | MTBI
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/11
Other Adverse Events (participants affected / at risk) | 0/15 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes